CLINICAL TRIAL: NCT00282945
Title: Analyzing Beta Cell Function Tests Over Time In Patients With Type 2 Diabetes Mellitus Randomized To Metformin Or Rosiglitazone
Brief Title: Beta Cell Function Tests Over Time In Patients With T2dm Randomized To Metformin Or Rosiglitazone
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: See statement in Detailed Description.
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: A9001289
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone; Metformin

INTERVENTIONS:
Drug: Rosiglitazone
Drug: Metformin

SUMMARY:
The purpose of this study is to determine whether markers of b-cell function can predict changes in B-cell function over time in patients with type 2 diabetes mellitus (T2DM) randomized to treatment with metformin or rosiglitazone.

DETAILED DESCRIPTION:
The study terminated on 17-Jul-07 due to concerns about long-term cardiovascular safety of Avandia and slow patient enrollment. There were no specific safety issues raised within the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with type diabetes mellitus (diagnosed via ADA criteria), newly diagnosed or treatment-naive (other than diet and exercise) and HbA1c range of 7 to 9%.
* 45-70 years of age.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (excluding untreated, asymptomatic, seasonal allergies).

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-01; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
This study will examine whether biomarkers of B-cell function measured early in the study (1, 3, and/or 6 months) will predict long-term changes in B-cell function (as represented by HOMA-B).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Israel (2):
  - Pfizer Investigational Site, Holon
  - Pfizer Investigational Site, Jerusalem

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001289&StudyName=Beta%20Cell%20Function%20Tests%20Over%20Time%20In%20Patients%20With%20T2dm%20Randomized%20To%20Metformin%20Or%20Rosiglitazone